CLINICAL TRIAL: NCT07084571
Title: Feasibility of Serial Multisite Image-Guided Biopsy To Study Breast Cancer Evolution
Acronym: FORTITUDE
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5876
Record Dates: First submitted 2025-07-02; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Triple Negative Breast Cancer
Keywords: Interventional Radiology
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples Blood samples Biological fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
FORTITUDE is a translational research study that aims to collect serial multi-site needle biopsy samples of tumour tissue and blood from metastatic breast cancer patients. Cancer biopsies are generally performed when cancer is diagnosed and are sometimes repeated when the cancer is suspected to have spread but this is not mandatory. However, studies have shown that cancers change with time and evolve to become resistant to therapy. The purpose of this study is to assess the feasibility of biopsies of multiple cancer sites across different time points during treatment and understand how cancers evolve and change throughout treatment. The findings of this study could pave the way for using cancer biopsies more frequently in the clinic to pick up changes in cancer behaviour that could influence treatment choice. The samples collected from this study will be used for molecular and genetic research to increase our understanding of how metastatic breast cancer changes during treatment and will enable us to develop new cancer treatments and new ways of monitoring response to cancer therapies.

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed cancer in women and is the second leading cause of female cancer death in the UK. Metastatic breast cancer has a historical five-year survival of 26% in England, although there is considerable variation by histology, with the poorest outcomes observed in patients with triple negative breast cancer (TNBC). Therapeutic approaches are chosen based on tumour clinical and pathological features, including oestrogen hormone receptor (ER) and human epidermal growth factor receptor 2 (HER2) status, however, patients with advanced disease almost inevitably develop therapy resistance and disease progression.

Next generation sequencing technologies have allowed us to understand the biology of breast cancer at a previously unprecedented depth. While the molecular landscape of early breast cancer has been extensively investigated, our understanding of the molecular basis of metastatic breast cancer remains more limited. In the clinic, metastatic breast cancer tissue is often biopsied once, from a single site, at the time of diagnosis. This biopsy sampling method is under-representative of the total disease burden and does not take into consideration the fact that metastatic disease is heterogeneous and evolves during the course of the disease.

The development of a method to serially sample multiple disease sites that is acceptable to patients will allow comprehensive evaluation of the heterogeneity of their disease and allow a deeper understanding of tumour heterogeneity, the mechanisms underlying treatment resistance as well as the biological processes governing metastatic behaviour. This will enable us to develop new cancer treatments and new ways of monitoring response to cancer therapies.

FORTITUDE will evaluate established standard of care biopsy techniques (fine needle biopsy and core needle biopsy) in a serial and multisite approach in patients with metastatic breast cancer or with locally advanced but inoperable breast cancer. Tumour tissue will be acquired at:

1. Baseline (mandatory), defined as:

   1. At diagnosis of locally advanced but inoperable breast cancer or metastatic disease OR
   2. In patients with established locally advanced but inoperable breast cancer or metastatic disease who require re-biopsy for clinical reasons
2. At every diagnosis of disease progression (optional)

No more than a total of four lesions will be biopsied in one sitting, with a maximum of three anatomical sites targeted (and no more than two solid organs). When tissue sampling is required as part of clinical care, patients will be invited to undergo additional serial multisite sampling. The sampling scheme will be repeated at subsequent relevant time points. This will be coupled with blood sampling when clinically indicated, including prior to each cycle of systemic therapy, and on disease progression. Furthermore, any cerebrospinal, ascitic and pleural fluid drained as part of clinical care can also be collected and profiled within this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced, inoperable breast cancer or metastatic breast cancer OR radiological evidence of metastatic disease with a high index of suspicion that this is a recurrence of a previously diagnosed breast cancer.
2. Be aged 18 years and over.
3. Have given written informed consent to participate.

Exclusion Criteria:

1. Metastatic disease limited to bones, without a soft tissue component.
2. Any bleeding disorders or anticoagulation that cannot be corrected and that would render the risk of biopsy unacceptable.
3. If the consultant physician involved in the care of the patient assesses and decides the risk of the biopsy procedures is significant, defined as greater than 1% risk of significant complication.
4. Eastern Cooperative Oncology Group performance status of 3 and higher.
5. Known chronic infectious disease (Hepatitis B and C, HIV) that may impact patient safety.
6. Presence of any psychological, familial or sociological condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic breast cancer or locally advanced, inoperable breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2040-04 (Estimated); Study Completion 2040-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having two or more tumour sites sampled in one procedural sitting when technically feasible | Through study completion, 15 years
Proportion of patients having longitudinal sampling in those progressing on treatment | Through study completion, 15 years
Proportion of patients willing to undergo multisite sampling again in the future if clinically required | Through study completion, 15 years

SECONDARY OUTCOMES:
Quantification of procedural complication rates | Through study completion, 15 years
Quantification of duration of biopsy procedures | Through study completion, 15 years
Accuracy of tumour biopsies | Through study completion, 15 years
  Accuracy may be defined as the successful identification of tumour tissue through biopsy, as confirmed by histopathology examination, or by other exploratory means such as using CT images to measure actual needle tip position compared to planning scans
Quantification of proportion of samples adequate for molecular profiling | Through study completion, 15 years
Number of clinically relevant molecular alterations detected using multisite, multiregion, and serial sampling | Through study completion, 15 years
  This outcome will assess whether the use of multisite (different anatomical locations), multiregion (multiple regions within a single tumor), and serial (longitudinal, across time points) sampling strategies increases the detection of clinically relevant molecular alterations, compared to standard single-site or single-timepoint sampling.
Characterisation of change in molecular phenotypes and genotypes between different regions in a single tumour | Through study completion, 15 years
Characterisation of change in molecular phenotypes and genotypes between different tumours across time | Through study completion, 15 years
Concordance and comparison of molecular alterations between liquid biopsies (blood, ascites, pleural fluid) and tumour needle biopsy samples | Through study completion, 15 years
Characterisation of molecular and imaging tumour profiles and correlation with clinical characteristics, treatment responses and patient outcomes | Through study completion, 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen-John Sammut, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, United Kingdom